CLINICAL TRIAL: NCT03932578
Title: Intrathecal Atropine Versus Intravenous Metoclopramide for Prevention of Nausea and Vomiting During Caesarian Section Under Spinal Anesthesia
Brief Title: Intrathecal Atropine vs IV Metoclopramide for Nausea & Vomiting During CS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MSA10
Record Dates: First submitted 2019-04-24; First posted 2019-04-30 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Nausea; Vomiting
Keywords: Cesarean section; Nausea and vomiting; Spinal Anesthesia
MeSH Terms: conditions — Nausea; Vomiting | interventions — Atropine; Metoclopramide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atropine group (Active Comparator): Patients will receive IV study solution which is 2 ml saline 0.9% as a placebo + intrathecal study solution which is a premised solution of 2.5 ml of 0.5% hyperbaric bupivacaine, 25 μg fentanyl and 100 μg of a 1 mg/ml preservative-free atropine sulfate solution
  Interventions: Drug: Atropine sulfate
- Metoclopramide group (Active Comparator): Patients in will receive IV study solution which is metoclopramide 10 mg in 2 ml + intrathecal study solution which is a premised solution of 2.5 ml of 0.5% hyperbaric bupivacaine, 25 μg fentanyl and 100 μg of preservative-free saline 0.9% as a placebo
  Interventions: Drug: Metoclopramide

INTERVENTIONS:
Drug: Atropine sulfate — Patients will receive intrathecal 100 μg of a 1 mg/ml preservative-free atropine sulfate solution
  Arms: Atropine group
Drug: Metoclopramide — Patients will receive IV metoclopramide 10 mg in 2 ml
  Arms: Metoclopramide group

SUMMARY:
The aim of this study is to evaluate the prophylactic use of low dose atropine and comparing it to metoclopramide for reducing intraoperative nausea and vomiting during cesarean section under spinal anesthesia

DETAILED DESCRIPTION:
Patients After obtaining the approval of the Mansoura Faculty of Medicine Institutional Research Board (MFM-IRB) and registration with ClinicalTrials.gov, this prospective double blind randomized study will be conducted in the next 6 months on 100 pregnant women undergoing elective CS in obstetric surgery unit in Mansoura University Hospital, Mansoura, Egypt. A written informed consent will be taken from each patient selected to participate before inclusion in the study.

Inclusion criteria Patients with ASA physical status class I or II; indications for CS other than fetal or maternal pathology and surgery scheduled for within 4 days of physiological term will be included in this study.

Exclusion criteria Patients with any of the following criteria will be excluded from the study: 1) age < 20 or > 35 years; 2) height < 150 or > 180 cm; 2) body mass index (BMI) >35 kg/m2; 4) active labor or emergency CS; 5) emesis gravidarum; 6) multifetal pregnancy; 7) fetal distress; 8) associated medical problem with pregnancy (as hypertension, diabetes mellitus, hepatic impairment or renal impairment);9) obstetric problem (as placenta previa or placental abruption); 10) contraindication for central neuraxial block; 11) history of adverse reaction to any study medication; 12) history of antiemetic drug use; or 13) refusal to undergo regional anesthesia.

Methods All patients participating in the study will be randomly divided into two groups; atropine group and metoclopramide group. The randomization will be simple and balanced (1:1) and will be carried out by a nurse through sealed, unlabeled, opaque envelopes containing computer-generated random numbers. The participants, caregivers and investigators will be blinded to group assignment. Patients in the atropine group will receive IV study solution which is 2 ml saline 0.9% as a placebo + intrathecal study solution which is a premised solution of 2.5 ml of 0.5% hyperbaric bupivacaine, 25 μg fentanyl and 100 μg of a 1 mg/ml preservative-free atropine sulfate solution. Patients in the metoclopramide group will receive IV study solution which is metoclopramide 10 mg in 2 ml + intrathecal study solution which is a premised solution of 2.5 ml of 0.5% hyperbaric bupivacaine, 25 μg fentanyl and 100 μg of preservative-free saline 0.9% as a placebo.

All participants will be instructed to stop oral intake 8 hours before surgery, but they will be allowed to drink moderate amounts of water and juices until 6 hours before surgery. Anesthesia protocol will be standardized in all patients. On arrival of the patient to operative theatre, intravenous (IV) cannula will be inserted and IV infusion of Ringer's acetate (8 ml/kg) will be given over about 20 minutes as a fluid preload before anesthesia. Patients will receive the IV study solution (according to their allocation) 15 minutes before start of anesthesia procedures. The spinal anesthesia will be performed in sitting position under strict aseptic condition. The anesthesia will be given at the level of L2-L3 or L3-L4 with a 25-gauge whit acre needle. Injections will be made using three separate syringes. Patients will be placed in a supine position immediately after the end of injections. A left lateral posture will be applied to all patients.

Sensory block will be assessed every 2 minute after intrathecal injection by using analgesia to pinprick in midclavicular line until achieving a stable level of sensory block. Surgery will be permitted after achieving T6 sensory block level. If the sensory level will not reach this level this case will be excluded from the study, and general anesthesia will be then given. Motor block will be assessed by using modified Bromage score (BS) in which, BS0 means no motor block; BS1 means inability to raise extended legs; BS2 means inability to flex knees; BS3 means inability to flex ankle joints. Complete motor block will be defined as BS3.

Heart rate, noninvasive arterial blood pressure and peripheral oxygen saturation (SpO2) measurements will be assessed in both groups preoperatively, during shifting and every 10 minutes intraoperatively. Hypotension will be defined as systolic blood pressure < 100 mmHg or > 30% decrease in baseline values. Bradycardia will be defined as heart rate < 60 bpm or a 20% drop in heart rate. Hypotension will be treated initially by bolus IV infusion of crystalloids (300 ml) then IV ephedrine 5 mg will be administered as needed. Bradycardia will be treated with fluids, positioning and ephedrine (up to 25 mg).If bradycardia does not resolve within seconds of treatment, IV atropine sulphate 0.5 mg will be given every 30 seconds until resolution. Patients who will receive IV atropine in addition to the study dose will be excluded from the study. After delivery, bradycardia will be only treated if hypotension is also present, or when the heart rate is <60 bpm.

Outcome measures The main outcome measure will be occurrence of IONV or PONV. Any IONV or PONV rating > 3 or spontaneous reporting of IONV or PONV by patients during scheduled interviews, as well as any clinical manifestations (retching or vomiting) and any requests for antiemetic medication will be considered as episodes of NV. Other outcome measures will be pain at rest, hypotension, bradycardia, shivering, pruritus, unexplained anxiety, xerostomia, photophobia, and the time of the first request for antiemetic drugs and analgesics and the number of requests until 12 h postoperatively.

Statistical analysis The statistical analysis will be performed using the IBM® SPSS® Statistics, version 20.0 for Windows. Continuous variables will be expressed as mean ± standard deviation (SD) and categorical variables will be expressed as frequencies and percentages. The normality distribution of continuous variables will be tested with the Kolmogorov-Smirnov and Shapiro-Wilk tests. Differences among continuous variables with normal distribution will be compared with the t-test while for continuous variables without normal distribution, non-parametric tests will be used and differences will be compared with the Mann-Whitney U-test. Differences between percentages will be compared with the Fisher's exact test. P values ≤ 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA physical status class I or II; indications for CS other than fetal or maternal pathology and surgery scheduled for within 4 days of physiological term will be included in this study

Exclusion Criteria:

* Height < 150 or > 180 cm
* Body mass index (BMI) >35 kg/m2
* Active labor or emergency CS
* Emesis gravidarum
* Multifetal pregnancy
* Fetal distress
* Associated medical problem with pregnancy (as hypertension, diabetes mellitus, hepatic impairment or renal impairment)
* Obstetric problem (as placenta previa or placental abruption)
* Contraindication for central neuraxial block
* History of adverse reaction to any study medication
* History of antiemetic drug use
* Refusal to undergo regional anesthesia

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-05 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Intraoperative nausea and vomiting (IONV) | During CS
  Spontaneous reporting of IONV by patients, as well as any clinical manifestations (retching or vomiting) and any requests for antiemetic medication will be considered as episodes of NV
Postoperative nausea and vomiting (PONV) | 12 hours after CS
  Spontaneous reporting of PONV by patients during scheduled interviews, as well as any clinical manifestations (retching or vomiting) and any requests for antiemetic medication will be considered as episodes of NV

SECONDARY OUTCOMES:
Time of requiring antiemetics | Until 12 hours postoperatively
  The time of the first request for antiemetic drugs
Number of requiring antiemetics | Until 12 hours postoperatively
  The number of requests for antiemetic drugs

CONTACTS AND LOCATIONS:
Overall Officials: Tamer Elmetwally, MD, Principal Investigator — Mansoura University; Mohamed S Abdelhafez, MD, Study Chair — Mansoura University
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication and forever
Access Criteria: Contact to corresponding author